CLINICAL TRIAL: NCT01091818
Title: A Prospective, Double-blind Study of Dexmedetomidine Versus Midazolam for Intensive Care Sedation of Children
Brief Title: Dexmedetomidine Versus Midazolam for Intensive Care Sedation of Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Johan Rader/Professor, University of Oslo
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: dexmedetmidazchildintsed
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Sedation
Keywords: To see if sedation with dexmedetomidine results in faster emergence after end of intensive care treatment in children; treatment
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- midazolam (Active Comparator)
  Interventions: Drug: Midazolam
- dexmedetomidin (Experimental)
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — Dexemedethomidine is given as major sedative drug
  Other Names: Midazolam is given as major sedative drug
  Arms: dexmedetomidin
Drug: Midazolam — Midazolam is given as major sedative drug
  Arms: midazolam

SUMMARY:
Dexmedetomidine will be tested against midazolam in a prospective, randomized, double-blind study of intensive care children, age 2-17 years.

The investigators' primary hypothesis is that time from end of medication to extubation will be shorter with dexmedetomidine sedation.

ELIGIBILITY:
Inclusion Criteria:

* informed consent from parents
* age between 2 and 18 years
* anticipated need of respirator treatment for more than 24 hrs
* included in study within 48 hrs of admission to intensive care unit (ICU)

Exclusion Criteria:

* severe, unstable circulatory failure
* severe intracranial or spinal trauma with circulatory instability
* sever bradycardia or atrioventricular (A-V) block
* liver failure
* less than 50% chance of anticipated survival
* known allergy to study drugs

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Time from end of sedation to extubation | 1-24 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Anesthesiology, Oslo University Hospital, Ullevaal, Oslo, Norway